CLINICAL TRIAL: NCT05326100
Title: Use of Virtual and Augmented Reality Devices in Vestibular Physical Therapy for mTBI
Acronym: VR4VPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Naval Health Research Center (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Pinata Sessoms, Research Biomedical Engineer, Naval Health Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2020-0332
Record Dates: First submitted 2022-03-03; First posted 2022-04-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Dysfunction of Vestibular System
Keywords: Virtual Reality; Augmented Reality; Vestibular Physical Therapy; Computer Assisted Rehabilitation Environment (CAREN); Head Mounted Display (HMD); Physical Therapy; MTBI; Servicemember; Vestibular Dysfunction
MeSH Terms: conditions — Brain Concussion | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Conventional Therapy (CPT) Group (Active Comparator): Each session will include vestibular exercises, customized to address the participant's symptoms of vestibular dysfunction and functional ability.
  Interventions: Other: Conventional Therapy (CPT)
- CAREN Group (Active Comparator): The CAREN group will undergo vestibular physical therapy that will include virtual environment (VE) applications on the CAREN.
  Interventions: Device: CAREN Therapy
- Augmented Reality (AR) Group (Experimental): The AR group will undergo vestibular physical therapy that will include VE applications on the AR HMD.
  Interventions: Device: Augmented Reality (AR) Therapy

INTERVENTIONS:
Other: Conventional Therapy (CPT) — The exercises may include traditional vestibulo-ocular reflex (VOR) exercises, cervical musculoskeletal exercises, somatosensory exercises, habituation, gait exercises, and aerobic conditioning. The treating PT will modify specific exercises as appropriate based on the participant's symptoms.
  Arms: Conventional Therapy (CPT) Group
Device: CAREN Therapy — The CAREN, an FDA-registered exempted Class I device, is a VR-based system which includes a six degree-of-freedom motion platform with an embedded, instrumented treadmill surrounded by an immersive 180-degree screen. The CAREN can display a variety of virtual environments (VEs), where the difficulty level and task requirements can be easily modified by the treating clinician to target patient-specific needs.
  Arms: CAREN Group
Device: Augmented Reality (AR) Therapy — AR head-mounted displays are designed to provide immersive virtual environments similar to the CAREN, but with the portability to be used in most outpatient clinical settings and potentially for at-home therapy as well as significantly reduced cost compared to the CAREN. AR devices have integrated eye-tracking and inertial measurement units (IMUs) which can be used to objectively quantify characteristics of eye, head and body movement.
  Arms: Augmented Reality (AR) Group

SUMMARY:
Rapidly evolving virtual reality (VR) and augmented reality (AR) technologies are being incorporated by many large-scale industries, and the medical field is no exception. One area that has gained significant attention in recent years is virtual rehabilitation which allows physical therapists to leverage state-of-the-art immersive virtual environments to uniquely address functional deficits in patients who are unresponsive to conventional treatment techniques. Advanced VR and AR technologies are now available in commercially available small-scale, mobile head-mounted displays which can be readily used in outpatient clinic settings and possibly at home.

The aim of this study is to determine whether advanced VR- and AR-based physical therapy improves functional status and reduces self-reported symptoms in individuals experiencing vestibular disorders secondary to mild traumatic brain injury (mTBI). Study participants will be randomized into treatment groups: 1) conventional therapy, 2) therapy performed using a large-scale VR system (the Computer Assisted Rehabilitation Environment or CAREN), 3) therapy performed using a mobile AR. Upon completion of treatment, groups will be compared to determine functional outcome improvements with respect to static and dynamic balance as well as reduction of vestibular symptoms.

DETAILED DESCRIPTION:
This protocol represents Phase 2 of a project that seeks to implement mobile AR-based technologies into vestibular physical therapy. The Phase 1 protocol (EIRB Number - NHRC.2019.0002) is ongoing and will compare outcomes from the AR-based HMD system (e.g., Magic Leap One) to the VR-based CAREN system. With validated instruments from Phase 1, this pilot prospective, three-armed randomized, interventional clinical trial seeks to incorporate advanced VR- and AR-based technologies as modalities in physical therapy for servicemembers (SMs) with mTBI who also experience vestibular dysfunction. The three arms are: 1) conventional vestibular physical therapy only (CPT), 2) CAREN only (CAREN), and 3) AR HMD only (AR).

Primary:

To determine whether advanced VR- and AR-based therapy, improves functional status and reduces self- reported symptoms in SMs with vestibular dysfunction and a history of mTBI.

Hypothesis: The investigators hypothesize that after completion of vestibular physical therapy, participants in the CAREN and AR groups will have better outcomes than those in the CPT group. In the CAREN and AR groups, the investigators anticipate greater improvements in static and dynamic balance, as measured by the Sensory Organization Test (SOT), Community Balance and Mobility Scale (CB&M), and Functional Gait Assessment (FGA), as well as decreased vestibular symptoms, as measured by the Dizziness Handicap Inventory (DHI) and Activity-Specific Balance Confidence Scale (ABC).

Secondary:

To determine whether participants in the advanced technology groups demonstrate similar clinical improvements following treatment.

Hypothesis: The investigators hypothesize that after completion of vestibular physical therapy, participants in the CAREN and AR groups will show similar improvements in static and dynamic balance as well as vestibular symptoms; essentially, the investigators believe the VR- and AR-based therapies will be comparable.

Tertiary:

To investigate the user experience associated with utilizing advanced technology for the treatment of vestibular dysfunction.

Hypothesis: The investigators hypothesize that participants in the AR group will have greater satisfaction than the CAREN group, as measured by higher scores on the User Satisfaction Evaluation Questionnaire (USEQ).

Exploratory:

Efforts from this study seek to gather information to justify further implementation of AR-based therapy (using HMDs) as well as the development and incorporation of additional military-relevant tasks, such as return-to-duty tasks and measures to be developed for future research efforts.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, active duty SMs between 18 and 65 years of age and enrolled in Defense Enrollment Eligibility Reporting System (DEERS)
* History of mTBI based on the Ohio State University Traumatic Brain Injury Identification (OSU TBI-ID)
* Require vestibular physical therapy as determined by a PT
* Normal or corrected vision based on the Snellen Eye Chart of at least 20/40
* Able to consistently follow verbal and written instructions and observe safety precautions
* Able to tolerate up to 60 minutes of physical therapy exercise, with breaks
* Able to ambulate with contact guard assistance or less, and to walk unassisted over ground or on a treadmill for 10 minutes at a time
* Able to tolerate wearing a full body safety harness
* Able to tolerate wearing a head mounted display weighing up to 3 pounds for up to 60 minutes

Exclusion Criteria:

* History of a moderate or severe TBI (OSU TBI-ID; or DVBIC TBI Screening Tool)
* Under care of a physician for a neurodegenerative diagnosis
* History of seizures or syncope
* Clinical determination of Benign Paroxysmal Positional Vertigo (BPPV)
* Diagnosis of any of the following visual impairments: field cuts, macular degeneration, retinal detachment, diplopia, limited peripheral or central vision, or require prism lenses
* Unable or unwilling to use contacts for corrected vision
* Require a medical device that can be affected by radio waves such as a pacemaker, defibrillator, or hearing devices (implantable or air conduction)
* Medications with significant sedating side effects that could impact safety (i.e., Phenobarbital, Ativan, etc.)
* Women who are more than 4 months pregnant may not participate in this study due to the effects advanced pregnancy can have on balance and vision. Note: Women who choose to participate will be informed up front that there are risks associated with pregnancy including decrements in postural control and falls. Additionally, changes in hormones, metabolism, fluid retention, and blood circulation during pregnancy can affect the eyes and eyesight. Women who become pregnant during the intervention should inform their PT immediately to determine if continued participation is possible.
* Concurrent participation, either clinically and/or as a part of another research study, in vestibular physical therapy and/or PTSD treatment
* Unable to consent for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Functional Assessments: Sensory Organization Test (SOT) | 6 weeks
  Assessment consisting of six different conditions used to measure balance and postural control. This test will be performed on the Neurocom Equitest Balance Manager and administered by a physical therapist. The first three conditions have a fixed surface, but the final three conditions are completed with a sway-referenced surface. The visual input is also changed between conditions, completed with eyes open or closed, or with either a fixed or sway referenced visual surroundings. The composite score, a weighted average of the six conditions, is able to distinguish between individuals that are healthy (higher composite scores) and those with balance deficits (lower composite scores). The test will take approximately 15 minutes to complete and will be administered at evaluation and re-evaluation.
Functional Assessments: Community Balance and Mobility Scale (CB&M) | 6 weeks
  Assessment used to evaluate the performance of 13 tasks for ambulatory individuals with TBI, and has been found to be valid and reliable, and sensitive in this population. Each task is scored on a scale of 0-5 based on the success of task completion, with a maximum score of 96. The tasks evaluated are unilateral stance, tandem walking, 180 degree tandem pivot, lateral foot scooting, hopping forward, crouch and walk, lateral dodging, walking and looking, running with controlled stop, forward to backward walking, walk, look and carry, and descending stairs. This will take approximately 20-30 min to complete and will be administered at evaluation and re-evaluation.
Functional Assessments: Functional Gait Assessment (FGA) | 6 weeks
  Assessment composed of 10 gait tasks, administered and scored on a 0-3 ordinal scale by a physical therapist. Scoring is based on the ability to walk over a level surface, change speed, walk while turning the head, walk and pivot, step over an obstacle (approximately 6" in height), walk with a narrow base of support (heel to toe), walk with eyes closed, walk backwards, and walk up steps, with a lower score indicating a higher degree of impairment. This will take approximately 5-10 minutes to complete and will be administered at evaluation and re-evaluation.
Vestibular Symptoms: Activity-Specific Balance Confidence Scale (ABC) | 6 weeks
  Questionnaire of self-reported balance confidence in daily activities developed to measure the psychological impact of balance impairment and/or falls. Participants score 16 items on a scale of 0% (no confidence) to 100% (total confidence) that they can perform the activity without losing balance. The ABC has been proven to be internally consistent, reliable, and valid. This will take approximately 5 minutes to complete and will be administered at evaluation and re-evaluation.
Vestibular Symptoms: Dizziness Handicap Inventory (DHI) | 6 weeks
  Evaluation of self-perceived handicapping of the effects imposed by dizziness. The DHI is constructed of 25 questionnaire items classified into three subgroups: physical (0-28 points), emotional (0-24 points), and functional (0-48 points). Answers are graded 0-4 with total score ranges from 0 to 100, 100 signifying the highest degree of impairment. The questionnaire has been validated and is sensitive to subtle balance deficits following mild TBI. This will take approximately 10 minutes to complete and will be administered at evaluation and re-evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Pinata Sessoms, PhD, Principal Investigator — Naval Health Research Center; Sarah Kruger, MS, Principal Investigator — Walter Reed National Military Medical Center; Kerry Rosen, PhD, Principal Investigator — Walter Reed National Military Medical Center
Locations (3):
- United States (3):
  - Naval Health Research Center, San Diego, California
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No